CLINICAL TRIAL: NCT05804630
Title: Efficacy and Safety of Articaine and Lidocaine in Extraction of Wisdom Teeth of Upper and Lower Jaws
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 202211014MINB
Record Dates: First submitted 2023-02-13; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-01

CONDITIONS: Wisdom Tooth; Dental Impaction
Keywords: Dental anesthesia; Lidocaine; Articaine; Wisdom tooth; Third molar; Impaction
MeSH Terms: conditions — Tooth, Impacted | interventions — Carticaine; Lidocaine

STUDY DESIGN:
Intervention Model Description: Split-mouth study design: one dental anesthetic agent at one side (left or right) of mouth and another agent at the other (left or right) side of mouth
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experiment 1, arm 1: Articaine infiltration anesthesia (Active Comparator): This arm aims to compare efficacy and safety of infiltration anesthesia of Articaine (Orabloc®) to block anesthesia of Lidocaine (Octocaine®). It would be a split-mouth study design. The patient in this arm would be randomly assigned to one anesthetic agent and technique at one side (left or right) of the wisdom tooth surgery first, and the other side (left or right) of wisdom tooth surgery would use the other anesthetic agent and technique accordingly.
  Interventions: Drug: Different dental anesthetic agents during wisdom tooth surgery (Orabloc®, Octocaine®, and Xylestesin-A®)
- Experiment 1, arm 2: Lidocaine block anesthesia (Active Comparator): This arm aims to compare efficacy and safety of infiltration anesthesia of Articaine (Orabloc®) to block anesthesia of Lidocaine (Octocaine®). It would be a split-mouth study design. The patient in this arm would be randomly assigned to one anesthetic agent and technique at one side (left or right) of the wisdom tooth surgery first, and the other side (left or right) of wisdom tooth surgery would use the other anesthetic agent and technique accordingly.
  Interventions: Drug: Different dental anesthetic agents during wisdom tooth surgery (Orabloc®, Octocaine®, and Xylestesin-A®)
- Experiment 2, arm 1: Lidocaine+1:100000 adrenaline block anesthesia (Active Comparator): This arm aims to compare efficacy and safety of block anesthesia of Lidocaine containing different concentration of epinephrine (adrenaline), i.e. Octocaine® (Lidocaine+1:100000 adrenaline) vs. Xylestesin-A® (Lidocaine+1:80000 adrenaline). It would be a split-mouth study design. The patients in this arm would be randomly assigned to one anesthetic agent at one side (left or right) of the wisdom tooth surgery first, and the other side (left or right) of wisdom tooth surgery would use the other anesthetic agent accordingly.
  Interventions: Drug: Different dental anesthetic agents during wisdom tooth surgery (Orabloc®, Octocaine®, and Xylestesin-A®)
- Experiment 2, arm 2: Lidocaine+1:80000 adrenaline block anesthesia (Active Comparator): This arm aims to compare efficacy and safety of block anesthesia of Lidocaine containing different concentration of epinephrine (adrenaline), i.e. Octocaine® (Lidocaine+1:100000 adrenaline) vs. Xylestesin-A® (Lidocaine+1:80000 adrenaline). It would be a split-mouth study design. The patients in this arm would be randomly assigned to one anesthetic agent at one side (left or right) of the wisdom tooth surgery first, and the other side (left or right) of wisdom tooth surgery would use the other anesthetic agent accordingly.
  Interventions: Drug: Different dental anesthetic agents during wisdom tooth surgery (Orabloc®, Octocaine®, and Xylestesin-A®)

INTERVENTIONS:
Drug: Different dental anesthetic agents during wisdom tooth surgery (Orabloc®, Octocaine®, and Xylestesin-A®) — As mentioned in arm/group descriptions. The amount of dental anesthetic agents used during the surgery will be tailored for patient according to their response, which will not exceed the recommended dosage described in the instruction of the product. The amount of the drug used during the surgery will be recorded.

SUMMARY:
Local anesthesia drugs and anesthesia technique play an imperative role in dental treatment. The purpose of this study was to compare the efficacy and safety of different dental local anesthetics drugs and brands in clinical use for the extraction of wisdom teeth.

DETAILED DESCRIPTION:
Local anesthesia drugs and anesthesia technique play an imperative role in dental treatment. They are widely used in oral and maxillofacial surgery, endodontic treatment, periodontal treatment, prosthetics and operative dentistry. They not only reduce the pain of the patient during the treatment, but also improve the comfort of the treatment. The most commonly used local anesthetics are Lidocaine and Articaine, whose efficacy and safety have been demonstrated in many literatures: fast-acting, effective in pain control, comfortable, relatively rare allergic reaction, few local and systemic adverse effects.

Among the above-mentioned drugs, Articaine is an anesthetic drug that has been developed and become popular in recent years. In the past, literature pointed out that due to the relationship between the drug concentration and structure of Articaine, its ability to penetrate into bone is better than that of Lidocaine. Some studies even believe that local infiltration with Articaine can replace block anesthesia with Lidocaine; which means, on the one hand, it is more comfortable during anesthesia. On the other hand, it can avoid the potential adverse effects of block anesthesia, such as: hematoma formation and systemic adverse effects caused by intravascular injection.

For exodontia surgery, a quite common surgery for general dentists and oral surgeons, the most commonly used anesthesia techniques are local infiltration and block anesthesia. The purpose of this study was to compare the efficacy and safety of different dental local anesthetics drugs and brands in clinical use for the extraction of impacted wisdom teeth. Three types of local anesthetics that have been widely used and proven safe were included:

1. Xylestesin-A® (1.7mL/cartridge contains 20mg/mL Lidocaine + 1:80,000 epinephrine)
2. Octocaine® (1.8mL/cartridge contains 20mg/mL Lidocaine + 1:100,000 epinephrine)
3. Orabloc® (1.8mL/cartridge contains 40mg/mL Articaine + 1:100,000 epinephrine)

This study will be a randomized split-mouth clinical study, and it will include 60 healthy adult patients aged between 20-60 years old, who are evaluated by a single surgeon to be suitable for extraction or odontectomy of their impacted third molars (upper or lower jaws) under local anesthesia. This study consists of two experiments. The above 60 patients will be randomly assigned to group 1 or 2, using different anesthetic drugs or anesthesia techniques:

1. Group 1: Octocaine® block vs. Xylestesin-A® block
2. Group 2: Orabloc® infiltration vs. Octocaine ® block

During the treatment, we will record the patient's subjective anesthesia onset time, the physician's objective anesthesia onset time, the patient's pain scale during surgery, comfort assessment, adverse reactions, postoperative paresthesia, etc. to evaluate the efficacy and safety of these drugs and anesthesia technique.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 20-60 years old
* Generally healthy or with well-controlled mild systemic diseases (such as well-controlled hypertension, diabetes, or hyperlipidemia)
* Bilateral wisdom teeth with similar difficulty of surgery(according to Pell and Gregory and Winter's classification), which are indicated for surgical removal under local anesthesia

Exclusion Criteria:

* Known or suspected allergy to amide-type local anesthetic agents
* With systemic contraindication for tooth extraction, such as poorly-controlled heart diseases or diabetes, and severe liver or kidney diseases. Patients with systolic blood pressure greater than 150 mmHg or less than 90 mmHg or diastolic blood pressure greater than 100 mmHg or less than 60 mmHg are also excluded
* With local contraindication for tooth extraction, such as previous irradiation to the surgical region, acute infection or cellulitis at the surgical region
* Patients during pregnancy or lactation
* Patients taking analgesic or sedatives in 24 hrs
* Intolerant of dental extraction surgery under local anesthesia due to anxiety, dentophobia, or pain

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Hemodynamic measures | Recorded immediate before local anesthesia, immediate after local anesthesia, 5 minutes after local anesthesia and immediate after surgery
  Including heart rate (HR)
Hemodynamic measures | Recorded immediate before local anesthesia, immediate after local anesthesia, 5 minutes after local anesthesia and immediate after surgery
  Blood pressure (Systolic pressure and diastolic pressure)
O2 saturation (SpO2) | Recorded immediate before local anesthesia, immediate after local anesthesia, 5 minutes after local anesthesia and immediate after surgery
  O2 saturation (SpO2)
Pain and satisfaction of the surgery | Recorded immediate after each dental extraction surgery
  Pain according to VAS (0-10) and satisfaction score (1-5, "1" being the least satisfactory and "5" being the most satisfactory)

SECONDARY OUTCOMES:
Adverse events of anesthesia | Recorded during and interview the patient immediate after each dental extraction surgery
  Such as headache, dizziness, nausea, vomiting, tachycardia, dyspnea, or post-operative neurosensory disturbance

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dentistry National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Liau FL, Kok SH, Lee JJ, Kuo RC, Hwang CR, Yang PJ, Lin CP, Kuo YS, Chang HH. Cardiovascular influence of dental anxiety during local anesthesia for tooth extraction. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2008 Jan;105(1):16-26. doi: 10.1016/j.tripleo.2007.03.015. Epub 2007 Jul 25. PMID 17656135
- [Background] Malamed SF, Gagnon S, Leblanc D. Efficacy of articaine: a new amide local anesthetic. J Am Dent Assoc. 2000 May;131(5):635-42. doi: 10.14219/jada.archive.2000.0237. PMID 10832257
- [Background] Mikesell P, Nusstein J, Reader A, Beck M, Weaver J. A comparison of articaine and lidocaine for inferior alveolar nerve blocks. J Endod. 2005 Apr;31(4):265-70. doi: 10.1097/01.don.0000140576.36513.cb. PMID 15793381
- [Background] Evans G, Nusstein J, Drum M, Reader A, Beck M. A prospective, randomized, double-blind comparison of articaine and lidocaine for maxillary infiltrations. J Endod. 2008 Apr;34(4):389-93. doi: 10.1016/j.joen.2008.01.004. Epub 2008 Feb 7. PMID 18358883
- [Background] Kanaa MD, Whitworth JM, Corbett IP, Meechan JG. Articaine and lidocaine mandibular buccal infiltration anesthesia: a prospective randomized double-blind cross-over study. J Endod. 2006 Apr;32(4):296-8. doi: 10.1016/j.joen.2005.09.016. Epub 2006 Feb 17. PMID 16554198
- [Background] Lai TN, Lin CP, Kok SH, Yang PJ, Kuo YS, Lan WH, Chang HH. Evaluation of mandibular block using a standardized method. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Oct;102(4):462-8. doi: 10.1016/j.tripleo.2005.12.003. Epub 2006 Jun 8. PMID 16997112